CLINICAL TRIAL: NCT00221988
Title: A Randomized, Double-Blind, Cross-over Study of the Cognitive and Mood Effects of KEPPRA (Levetiracetam) Tablets in Healthy Older Adults.
Brief Title: Effects of Keppra on Thinking, Emotions, and Balance in Elderly Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Michael Schoenberg, Ignacio Pita, Kyra Dawson (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UCB MRS001; UHC 06-04-52
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Epilepsy
Keywords: Elderly; Epilepsy; Cognition; Health Outcome
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam (Keppra)

SUMMARY:
Epilepsy is a common disorder with an incidence of about 6 per 1000. The incidence progressively increases above age 50. By age 75, the incidence is two to three fold compared with any age group. Unfortunately, older individuals are especially at risk to incur significant side effects to anti-epileptic drugs. A newer anti-epileptic drug may markedly improve seizure management in older individuals as it is removed by the kidneys and not the liver and does not interact with other medications. We expect it to be tolerated well in terms of effects on memory, thinking,balance, and walking. The current study assesses the side effects of levetiracetam in healthy volunteers aged 65 to 80. Use of healthy volunteers eliminates the effects of seizures on the outcome.

DETAILED DESCRIPTION:
III. INTRODUCTION:

Background Antiepileptic Drugs And Cognitive Dysfunction Epilepsy is the most common debilitating neurologic disorder, with a prevalence of about 6/1000 in the general population (Hauser and Hesdorffer, 1990). Along with the disabling psychosocial and physical disadvantages that accompany epilepsy, medication concerns are frequently reported (Gilliam F et al. 1997). The majority of adverse events related to medications pertain to cognition (Baker GA et al. 1997).

A variety of factors contribute to cognitive dysfunction in persons with epilepsy, one of which is treatment with antiepileptic drugs (AEDs). The effects of AEDs appear to display a dose dependent relationship to cognitive functioning. Even more striking adverse effects on cognition are found as a result of AED polytherapy. Evaluation of the cognitive effects of AEDs in patients with epilepsy can easily be confounded by seizure effects, underlying cerebral injury, genetic, factors, and chronic impact of living with seizures. To limit the confounding cognitive effects of epilepsy, investigators have examined the cognitive effects of AEDs in healthy volunteers. Meador et al. (1995) have presented data demonstrating mild untoward effects of three common first line AEDs in a group of young healthy adults employing a randomized, double-blind, incomplete block crossover design. More than one-half of the neurocognitive dependent variables exhibited AED effects when compared with non-drug baselines. Studies of newer drugs have shown variable impairment with gabapentin and lamotrigine showing less impairment compared to the older, first-line drugs and to topiramate.

Epilepsy In The Elderly The incidence of epilepsy increases as age advances beyond 50. Indeed there is a two- to three-fold increase above the age of 75 years compared with any other age group (Ramsay et al. 2004). This special population is at increased risk for development of adverse events related to AED treatment as they are likely to have multiple medical conditions, take numerous concomitant medications, have different metabolic characteristics, and are more likely to suffer from neurologic conditions such as stroke and dementia. The elderly are more susceptible to cognitive impairment by AEDs. However, little is known of factors affecting health-related quality of life in senior adults with epilepsy (Martin et al., 2003)6. All older AEDs have clear pharmacokinetic disadvantages as they are liver metabolized with many known drug interactions.

Levetiractam Levetiracetam was approved by the FDA in 1999 for the treatment of epilepsy. Levetiracetam was shown to be an effective pharmacologic treatment for refractory partial seizures in a number of large multicenter clinical trials (French, et al., 2001; Cramer et al., 2003; Morrell et al., 2003). The pharmacokinetic profile of levetiracetam has particular advantages over other anti-epileptic drugs. Pharmacologic advantages include low protein binding, renal clearance, and an absence of drug interactions (Perucca and Johannessen, 2003.).

For the older patient with epilepsy, levetiracetam is likely to offer an excellent alternative to other AEDs that are known to interact with other medications. Levetiracetam has performed favorably in adults with epilepsy (Ben-Menachem & Gilland, 2003; Morrell et al., 2003). The efficacy of levetiracetam has been demonstrated for epilepsy in older adults (Cramer et al. 2003; Kraemer & Edrich, 2001).

Clinical experience suggests that Levetiracetam is a well-tolerated medication with minimal cognitive or sedative effects. Levetiracetam is a structural analogue of piracetam, a drug used as a nootropic (cognitive enhancing) agent in Europe. However, a recent placebo-controlled study of adjunctive levetiracetam therapy for intractable complex partial seizures showed several CNS adverse events more common than placebo, including somnolence, asthenia, and dizziness (Morrell et al., 2003). The occurrence of these specific cognitive adverse events were relatively modest ranging from one to seven per cent relative to placebo. Data detailing the cognitive and mood profile of levetiracetam in healthy older adults are limited. Kraemer and Edrich (2003) using pooled clinical trial data found no differences in the incidence of central nervous system events between elderly patients and younger adults in a large clinical trial. Similarly , the KEEPER trial found no difference in frequency of side effects to levetiracetam in younger verses adults over 65 (range 65 to>85) . The KEEPER trial was a phase IV study that has limited interpretability as it was open label (Ferrendelli et al., 2003). Clinical experience has been consistent in showing good tolerability in the elderly (French 2001 ;Cramer et al 2003a; Ferrendelli et al, 2003 ; Pryor and Ramsay, 2003 ; Ramsay et al,2003 ; Werz et al 2003 ; Alsaadi et al 2004). However, the neurocognitive and mood effects of levetiracetam in older adults have not yet been documented in well designed trials to specifically address this issue.

Studies have demonstrated similar seizure-free rates for the second generation AEDs, with the main difference being their side effect profile. Evidenced based medicine requires data to support prescription practices, and we hypothesize that the current data will provide support for the use of levetiracetam in older adults with epilepsy. We predict no significant effects of the study drug on cognition.

IV. STUDY OBJECTIVES AND ENDPOINTS Objective The primary objective of this study is to compare the effects of levetiracetam to placebo on neuropsychological and mood function in elderly healthy volunteers.

Study Endpoints

* Neuropsychological evaluations of cognitive function, behavioral responses, speech, and mood (See Appendix 1)
* Early discontinuation for adverse events V. STUDY DESIGN General Description This is a randomized, double-blind, placebo controlled, crossover study of levetiracetam in healthy older adults. The study is divided into 6 phases, which will occur over a total of 14 weeks: Screen (-2 weeks), Randomization (0 weeks), First Drug Treatment Period (4 weeks), Washout (2 weeks), Second Drug Treatment Period (4 weeks), and Post-Treatment (2 weeks) (Appendix 2). Each Drug Treatment Period is further divided into the Titration, Maintenance, and Taper Phases. Following Screening, subjects will be randomized (1:1) to receive either levetiracetam or placebo the First Drug Treatment Period. After completion of this phase and the subsequent Washout, subjects will receive the alternate therapy in the Second Drug Treatment Period.

Neuropsychological testing will be performed at screening, baseline, and during each maintenance phase. Each neuropsychological testing involves about two hours of pen and paper testing. A complete list of tests is given in Appendix 1.

Enrollment will occur at University Hospitals of Cleveland, Department of Neurology.

Study Population Inclusion Criteria

A subject will be eligible for inclusion in this study only if all of the following criteria apply. A subject must:

1. Provide a copy of their medical records from a primary care physician for the past year to assist in establishing the patient's current health status. The study physician will review PCP medical records to assure participants meet the study inclusion/exclusion criteria.
2. Be a healthy adult age 65 to 80 years old. Healthy subjects are defined as individuals who are free from significant cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, neurological and psychiatric disease as determined by history and physical examination.
3. Be, in the investigator's opinion, compliant, able to follow the investigator's instructions and visit the clinic on schedule, cooperative and reliable.
4. Subjects must score within -1.0 standard deviations of the mean performance of healthy individuals on the neuropsychological tests at screen (week -2). Subjects must have a reading equivalency of 8th grade. Participants must also have a MMSE score of 28. (Bravo & Herbert, 1997; Crum et al., 1993). Finally, participants must score a 45 or better on the Berg Balance Test at screening (week -2) to be included in the study.
5. Sign an informed consent.
6. For participants living alone, provide the name and number of at least one friend or family member that study personnel may contact in the unlikely event that study personnel are unable to contact the patient by phone past 48 hours of a scheduled phone contact time which was not planned.

Exclusion Criteria

A subject will not be eligible for inclusion in this study if any of the following criteria apply. A subject must not:

1. Have a history of any type of epilepsy.
2. Be taking any concomitant medications that are or any concomitant medications that may alter cognitive function or mood.
3. Have a current or past history of drug or alcohol abuse or dependence. Have a positive urine toxicology test at screen.
4. Have a history and clinical finding of a progressive encephalopathy including CNS tumors of all types.
5. Have a serious illness in the past month that may confound the interpretation of study results.
6. Be on anticoagulation with warfarin.
7. Have experienced a prior adverse reaction or hypersensitivity to either study medication or to related compounds.
8. Be currently participating in another clinical study in which the subject will be exposed to an investigational or a non-investigational drug or device.

Procedures to be performed and visit schedule Screening Clinic Visit 1(Visit 1, week -2): At screen, participating subjects will sign informed consent. Subjects will undergo exam to determine whether they qualify for participation in the study. Examination will include a complete physical and neurological examination, vital signs, neuropsychological assessment, MMSE, and Berg Balance Test. Neuropsychological assessment will require about 2 hours of pen and paper testing. Participants must score within -1.0 SD of the mean performance of age- and education-matched peers on each neuropsychological test. Participants must also not present on the physical or neurological exam with any exclusionary criteria Participants that meet the screening criteria will be invited back for the baseline visit (week 0). Subjects will be asked to bring with them at the baseline visit their medical records from their primary care physician and signed releases for their medical records will be obtained.

Randomization (week 0): Subjects will be randomized to receive either levetiracetam or placebo.

Baseline - Clinic Visit 2 (Visit 2, week 1): medical history, comprehensive physical and neurological examination, vital signs. Neuropsychological assessment will be completed. This involves pen and paper testing over about two hours. Laboratory evaluation will be performed including complete blood count, basic metabolic sceen including creatinine, hepatic function, coagulation parameters, and urine toxicology screen.

Study Drugs and Dosages KEPPRA (levetiracetam) 500 mg scored tablets will be supplied with matching placebo tablets. The dosage of levetiracetam will be about 1000 mg per day to be consistent with clinical experience with the elderly.

Titration During the Titration Phase of each Drug Treatment Period, doses of levetiracetam (or placebo) will be started at 250 mg twice a day (500 mg total daily dose) and increased over a period of two weeks to a target maintenance dose of 1000mg/day in divided dose, according to the dosing schedule outlined in the table that follows (Appendix 2). Upon achieving the target maintenance dose, subjects will receive this dose for one week during the Maintenance Phase. Following the Maintenance Phase, study drug will be tapered off over a period of one week and maintained off drug for one week (weeks 6 through 7) (washout period). The second treatment period will then begin (6 weeks).

Clinic Visit 3 (week 5) will occur at the end of the drug maintenance phase of the first Drug Treatment Period and include neurological examination, vital signs, and blood draw for drug serum concentration requiring about 60 minutes. Visit 2 will also include neuropsychological testing taking about two hours.

Clinic Visit 4 (week 7 - baseline 2) will occur at the end of the first drug washout and will involve a neurological and physical examination taking about 45-60 minutes. Subjects will complete Neuropsychological Assessment. Participants will then begin the second treatment phase.

Clinic Visit 5 (week 11) will occur at the end of the drug maintenance phase of the second drug treatment period and will also include neurological examination, vital signs, and blood draw for drug serum concentration taking about 60 minutes. Visit 5 will also include neuropsychological testing taking about two hours.

Clinic Visit 6 (Final visit, week 13): will occur after washout of the second drug and will again involve comprehensive physical and neurologic examination taking 45 to 60 minutes.

Phone calls will be made weeks 2, 3, 4, 6, 8, 9, and 12 to check on medication use and side effects for study participants that have a spouse or caregiver at home. Participants that report that they live alone will be called 3 times weekly during the study period (e.g., Monday, Wednesday, Friday).

VII. DATA ANALYSIS

A power analysis was conducted to determine the minimum sample size needed to detect changes on neuropsychological test scores with a formula for repeated measures of continuous data:

Although the within subject standard deviation (the standard deviation of repeated observations in the same individual) is unknown for studies with levetiracetam, data from similar research with anti-epileptic medications and published normative data for these tests suggests the within subject standard deviation varies from a standardized 0.1 to 0.6 units. A minimum power of 0.80 ( A minimum detectable difference in neuropsychological tests scores was set at a 0.5 units (a half a standard deviation in change for a neuropsychological test score). A standardized measure of mean difference was selected as the raw scores of neuropsychological instruments vary, and converting raw scores to standard scores allow all test scores to be compared using a common metric. Based on a two-tailed significance of 0.05, the minimum N needed is 18 subjects. With 20 participants, assuming a within subject standard deviation of 0.5 units, the minimum detectable difference will be 0.467 standard deviation units (slightly less than a ½ a standard deviation of change). It should be noted that for several neuropsychological tests the within subject change is less than 0.2 SD units. With a smaller within subject SD, and using the same parameters above, N = 20 yields a minimum detectable difference of 0.187 standard deviation units (small effect size). The change in neuropsychological measures found in other antiepileptic medications (e.g., carbamazepine and topiramate) has been from 0.2 to 2.5 units (e.g., Meador et al., 2001).

To obtain 20 completed subjects, experience from previous studies demonstrates a 50% dropout rate. Therefore, approximately 40 subjects will need to be enrolled to achieve the 20 completed participants for this study.

Analyses will be conducted on both intent-to-treat and per-protocol. Any subject who is valuable for the safety analysis that also has baseline and end of drug treatment period neuropsychological data available for each of the two drug periods will be evaluated for the intent-to-treat analyses of the parameters of interest. Mood and neuropsychological data will undergo analysis of variance (MANOVA) appropriate for a two-period crossover study. Alternative forms will be used when available. To compensate for practice effects and evaluate for measurement error, baseline will be defined as the average of the evaluations conducted at pre-treatment baseline and the post-treatment period (week 12).18 Subjects who discontinue prematurely will be tested two weeks after withdrawing. This will be considered the post-treatment period for these subjects.

VIII. Risks and Benefit There is no benefit to participating in this study. In the pivotal trials 15 % receiving Levetiracetam discontinued the study compared to 11.6% receiving placebo. Levetiracetam has reported only non-serious, reversible side effects. The most common significant side effect of levetiracetam is somnolence (i.e., lethargy), asthenia, infection, dizziness, and unsteady gait. Less common side effects include thinking abnormalities, memory problems, anxiety, depression, agitation, vertigo, and paresthesias. Rarely, levetiracetam has been associated with psychotic disturbance that resolved after treatment was discontinued (0.7%). The adverse event profile of levetiracetam is generally less than that to other medications such as lamotrigine, topiramate, phenytoin, carbamazepine, and bactrim. All study medication should be discontinued at the first sign of hallucinations.

VIII. Compensation. Subjects will be compensated for their time and inconvenience. Reimbursement assumes that a subject will invest about 14 hours over the three months of the study not including travel time. This is a significant imposition as we expect most volunteers to be gainfully employed. They will also be undergoing three blood draws and have the inconvenience of taking medications for almost two months. The compensation will be prorated to the amount of testing completed: $50 for screening visit, $200 for completing visit 3 (first treatment arm), $275 is given at visit 5 for completing the study. The maximal reimbursement is $525. Payment will be made at the end of participation in the study. Based on the subject volunteering 14 hours of their time, not including travel time, this equates to $37.50 per hour. This participation reimbursement rate is similar to the reimbursement rate of similar studies conducted at this institution and is also mirrored at other similar academic medical centers.

IX. Volunteer Recruitment and Confidentiality. Advertisements in the form of flyers (Appendix 3) will be distributed around University Hospital and Case Western Reserve University and in the hospital weekly flyer "Monday Morning". Volunteers face no harm to grades, job status, promotion or evaluation by participating or by withdrawing. Individuals within the Neurology Department will be excluded. Information will be confidential.

X. REFERENCES

1. Alsaadi, TM, Koopman, S, Apperson, M, Farias, S. Levetiracetam monotherapy for elderly patients with epilepsy. Seizure 2004;13(1):58-60.
2. Baker GA , Jacoby A, Buck D, Stalgis, C, Monnet, D. Quality of Life of people with epilepsy: a European study. Epilepsia 1997; 38:353-362.
3. Ben-Menachem E., & Gilland E. Efficacy and tolerability of levetiracetam during 1-year follow-up in patients with refractory epilepsy. Seizure 2003; 61:704-706.
4. Bravo G, & Herbert R. Age- and education-specific reference values for the Mini-mental and Modified Mini-Mental State Examinations derived from a non-demented elderly population. Intr J Geriatric Psychiatry 1997;12:1008-1018.
5. Cramer, JA, Leppik, IE, De Rue, K., Edrich, P., & Kraemer, G. Tolerability of levetiracetam in elderly patients with CNS disorders. Epilepsy Research 2003(a); 56:135-145.
6. Cramer JA., Katrie DR., Devinsky O., Edrich P., Trimble MR. A systematic review of the behavioral effects in levetiracetam in adults with epilepsy, cognitive disorders, or an anxiety disorder during clinical trials. Epilepsy Behav 2003(b); 4:124-132.French J., Edrich P., Cramer JA. (A systematic review of the safety profile of levetiracetam: A new antiepileptic drug. Epilepsy Res 2001; 47; 77-90.
7. Crum RM, Anthony JC, Bassett SS, Folstein MF. Population-based norms for the Mini-Mental State Exam by age and education level. Journal of the American Medical Association 1993, 269: 2389.
8. Ferrendelli J., French J., Leppik I., Morrell M., Herbeuval A., Han J., et al. Use of levetiracetam in a population of patients aged 65 years and older: A subset analysis of the KEEPERTM trial. Epilepsy Behav 2003;4:702-709.
9. Hauser, W.A., and Hesdorffer, D.C. Epilepsy: Frequency, causes, and consequences.

   New York: Demos Publications, 1990; 1-51.
10. Kraemer G., Edrich P. Levetiracetam in elderly patients with epilspsy [abstract]. Epilepsia 2001;42(Suppl 7):142-3.
11. Martin R., Vogtle L., Gilliam F., and Faught E. Health related quality of life in senior adults with epilepsy: what we know from randomized clinical trials and suggestions for future research. Epilepsy and Behavior 2003, 4:626-634.
12. Meador, K.J., Loring, D.W., Moore E.E., Thompson, W.A., Nichols, M.E., Oberzan, R.E., Durkin, M.W., Gallagher, B.B., and King D.W. Comparative cognitive effects of phenobarbital, phenytoin, and valproate in healthy adults. Neurology 1995; 45:1494-1499.
13. Meador, KJ, Loring, DW, Ray, PG, Murro, AM, King, DW, Perrine, KR, Vazquez, BR, Kiobasa, T. Differential cognitive and behavioral effects of carbamazepine and lamotrigine. Neurology 2001;56: 1177-1182.
14. Meador, KJ., Loring, DW., Werz, MA., Ray, PG., Schoenberg, MR., Ogrocki, P., & Kaul-Gupta, R. Perceived Preference for Lamotrigine or Topiramate: Correlation with self-report inventories and neuropsycholotgical testing. Poster presented at the 56th Annual Meeting of the American Academy of Neurology, San Francisco, CA, April 2004.
15. Morrell M., Leppik I., French J., Ferrendelli J., Han J., Magnus L. The KEEPERTM trial: Levetiracetam adjunctive treatment of partial-onset seizures in an open-label community-based study [published corrigendum appears in Epilepsy Res 2003; 56:209-210. Epilepsy Res 2003;54:153-61.
16. Perucca E and Johannessen SI. The ideal pharmacokinetic properties of an antiepileptic drug: how close does Levetiracetam come? Epileptic Disorders 2003, 5(suppl1):S17-S26.
17. Pryor FM, Ramsay RE, Keppra monotherapy in the elderly and in primary generalized epilepsy. 2003;44 suppl 9:270.
18. Ramsay et al. Evaluation of epilepsy in elderly subjects. Epilepsia 2004; 45 (Suppl 9): 16-21.
19. Ramsay, RE, Rowan, AJ, Pryor FM, Collins, JF. Treatment of seizures in the elderly: final analysis form DVA cooperative study #428. Epilepsia 2003;44 (suppl 9):170.
20. Werz, MA, Lang, P, Rienzo, T. Levetiracetam therapy for epilepsy: use and tolerability in the elderly. Epilepsia 2003;44 (suppl 9:280) (2.307).

ELIGIBILITY:
Inclusion Criteria:

* Study Population Inclusion Criteria

A subject will be eligible for inclusion in this study only if all of the following criteria apply. A subject must:

1. Provide a copy of their medical records from a primary care physician for the past year to assist in establishing the patient's current health status. The study physician will review PCP medical records to assure participants meet the study inclusion/exclusion criteria.
2. Be a healthy adult age 65 to 80 years old. Healthy subjects are defined as individuals who are free from significant cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, neurological and psychiatric disease as determined by history and physical examination.
3. Be, in the investigator's opinion, compliant, able to follow the investigator's instructions and visit the clinic on schedule, cooperative and reliable.
4. Subjects must score within -1.0 standard deviations of the mean performance of healthy individuals on the neuropsychological tests at screen (week -2). Subjects must have a reading equivalency of 8th grade. Participants must also have a MMSE score of 28. (Bravo & Herbert, 1997; Crum et al., 1993). Finally, participants must score a 45 or better on the Berg Balance Test at screening (week -2) to be included in the study.
5. Sign an informed consent.
6. For participants living alone, provide the name and number of at least one friend or family member that study personnel may contact in the unlikely event that study personnel are unable to contact the patient by phone past 48 hours of a scheduled phone contact time which was not planned.

Exclusion Criteria:

Exclusion Criteria

A subject will not be eligible for inclusion in this study if any of the following criteria apply. A subject must not:

1. Have a history of any type of epilepsy.
2. Be taking any concomitant medications that are or any concomitant medications that may alter cognitive function or mood.
3. Have a current or past history of drug or alcohol abuse or dependence. Have a positive urine toxicology test at screen.
4. Have a history and clinical finding of a progressive encephalopathy including CNS tumors of all types.
5. Have a serious illness in the past month that may confound the interpretation of study results.
6. Be on anticoagulation with warfarin.
7. Have experienced a prior adverse reaction or hypersensitivity to either study medication or to related compounds.
8. Be currently participating in another clinical study in which the subject will be exposed to an investigational or a non-investigational drug or device.

   -

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-03 (Actual); Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Objective Neuropsyhological testing
Subjective Behavioral Measures
Balance Measures

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann Werz, M.D., Ph.D., Principal Investigator — University Hospitals Cleveland Medical Center; Mike R Schoenberg, Ph.D., Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States